CLINICAL TRIAL: NCT05136118
Title: Transversus Abdominis Plane Block: Ultra-sound Guided Versus the Modified Surgeon Assisted Approaches for Post-operative Analgesia Following Cesarean Section
Brief Title: Transversus Abdominis Plane Block for Post-operative Analgesia Following Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor of Anesthesia, Intensive care and Pain Management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R 86/2021
Record Dates: First submitted 2021-10-08; First posted 2021-11-29 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Analgesia
Keywords: post-operative analgesia; Transversus Abdominis Plane Block
MeSH Terms: conditions — Agnosia | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MS (Active Comparator): The modified surgeon assisted approach for TAPB Before the closure of the peritoneum, TAPB will be performed; at the level of the umbilicus 8 to 10cms from the midline bilaterally. A sterile 100-mm 22-G insulated needle will be inserted perpendicular to the skin slightly directed towards the ipsilateral anterior superior iliac spine. After feeling the 2 pops of the external and the internal oblique aponeurosis by the anesthesiologist, the surgeon will confirm proper needle placement by his hand inside the abdominal cavity. The LA will be injected after negative aspiration and a bleb will be palpated by the surgeon as the injection continues. The same procedure will be repeated on the other side.
  Interventions: Procedure: TAPB
- Group US (Active Comparator): The ultra-sound guided approach for TAPB. After abdominal wall closure, the linear probe of the ultra- sound will be placed perpendicular to the skin at the mid-axillary line between the iliac crest and the costal margin; the TAP will be located between the internal oblique and the transversus abdominis muscle. A sterile 100-mm 22-G insulated needle will be inserted perpendicular to the skin and the 2 pops of the external and the internal oblique aponeurosis will be also felt. The LA will be injected after negative aspiration and its spread in the plane will be observed. The same procedure will be repeated on the other side.
  Interventions: Procedure: TAPB

INTERVENTIONS:
Procedure: TAPB — TAPB will be given to parturients whether by the modified surgeon assisted approach or by the ultra-sound guided approach.

SUMMARY:
Postpartum analgesia is a common concern after Cesarean Section (CS). The quality of postoperative recovery is improved by opioid sparing pain control approaches. The transversus abdominis plane block (TAPB) is an effective technique for postpartum analgesia after cesarean section. Pregnancy results in thinning of the internal oblique aponeurosis; with increased incidence of missing the second pop to reach the transversus abdominis plane (TAP). The classic blind approach to the TAP is associated with several complications; so, it has been largely replaced by the ultrasound-guided approach to the TAP. The ultrasound-guided approach to the TAPB was first described by Hebbart and his colleagues in 2007.Ultrasound-guided TAPB improves the success of the block, reduces the volume of local anesthetic used and prevents the potential injury of adjacent structures.

Surgical approach to the TAPB was also described, it is a quick and easy approach of establishing a reliable block. The surgeon performs an intra-abdominal approach to the TAPB; by which asepsis is easily attained, visible and tactile confirmation of correct needle placement may be achieved with no risk of damage to the viscera but care must be given to avoid injury of the inferior epigastric vessels.

DETAILED DESCRIPTION:
Compare the Transversus Abdominis Plane Block via the modified surgeon assisted approach (Study group), to the ultra-sound guided approach (Control group); as regards the post-operative analgesia following Cesarean Section.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and ∏
* primigravidas
* aged 21-40 years
* BMI ˂ 40
* body weight ˃ 60 kg
* singleton pregnancy
* gestational age of ≥37 weeks
* undergoing elective caesarean section under spinal anesthesia.

Exclusion Criteria:

* Parturient refusal
* parturient with a BMI > 40
* body weight < 60 kg
* ASA physical status ≥ III
* known local anesthetic (LA) allergy •contraindications to spinal anesthesia
* parturients who received analgesics in the past 24 hours
* infection at the site of the block.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 308 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Time to rescue analgesia | 6 months
  the time from the end of surgery until the first parturient's request for analgesia

SECONDARY OUTCOMES:
Efficacy of the modified surgeon assisted approach for TAPB on postoperative analgesia | 6 months
  assessment of pain intensity at rest and on passive flexion of the hip and knee by the Numeric Pain Rating Score (NPRS) from 0 = no pain to 10 = worst pain. Assessment will be done at 2, 6, 12 and 24h postoperative.
Number of parturients requiring postoperative analgesia | 6 months
  defined as pethidine needed by each parturient in the 24 hours postoperative period
Total dose of pethidine given | 6 months
  defined as pethidine needed by each parturient in the 24 hours postoperative period
Time to the parturient's first ambulation | 6 months
  the time to start of each parturient movement in the 24 hours postoperative period
The analgesic satisfaction 24 hours after operation | 6 months
  parturients will be asked to report their satisfaction with pain management, assessed as 0 = weak, 1 = medium, 2 = good, 3 = very good, and 4 = excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No